CLINICAL TRIAL: NCT00343408
Title: A Phase I, Open-Label, Dose-Seeking Study of AZD2171 Given Daily Orally in Combination With Selected Standard Chemotherapy Regimens (CT) in Patients With Advanced Incurable Non-Small Cell Lung Cancer (NSCLC) or Colorectal Cancer
Brief Title: AZD2171 and Standard Combination Chemotherapy in Advanced Non-Small Cell Lung Cancer or Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I175; CAN-NCIC-IND175 (Other: PDQ); CDR0000481443 (Other: PDQ)
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer; Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent colon cancer; stage III colon cancer; stage IV colon cancer; recurrent rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Colonic Neoplasms; Rectal Neoplasms | interventions — cediranib; Cisplatin; Fluorouracil; Gemcitabine; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: cediranib maleate
Drug: cisplatin
Drug: fluorouracil
Drug: gemcitabine hydrochloride
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: AZD2171 may stop the growth of tumor cells by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving AZD2171 together with standard combination chemotherapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of AZD2171 when given together with standard combination chemotherapy in treating patients with advanced non-small cell lung cancer (NSCLC) or colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the recommended phase II dose of AZD2171 when administered with standard combination chemotherapy in patients with advanced non-small cell lung cancer or colorectal cancer.
* Determine the safety, tolerability, toxicity profile, dose-limiting toxicities, and pharmacokinetic profile of this treatment regimen.
* Assess the antitumor activity of this treatment regimen in patients with measurable disease.
* Correlate the toxicity profile with pharmacokinetics.

OUTLINE: This is a multicenter, open-label, dose-escalation study of AZD2171. Patients are assigned to 1 of 2 treatment groups according to disease.

* Group 1 (non-small cell lung cancer): Patients receive gemcitabine hydrochloride IV on days 1 and 8 and cisplatin IV on day 1. Patients also receive oral AZD2171 once daily beginning on day 2. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
* Group 2 (colorectal cancer): Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours on days 1 and 2. Patients also receive oral AZD2171 once daily beginning on day 3. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.

In both groups, cohorts of 3-6 patients receive escalating doses of AZD2171 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of 1 of the following:

  * Non-small cell lung cancer (NSCLC), meeting 1 of the following criteria:

    * Stage IIIB disease

      * No pleural effusion and not a candidate for a combined modality treatment
    * Stage IV disease
    * Local or metastatic failure after surgery and/or radiotherapy
  * Colorectal cancer (CRC)

    * Advanced and/or metastatic disease
    * Suitable for first-line therapy with oxaliplatin, leucovorin calcium, and fluorouracil (FOLFOX-6)
* Clinically or radiologically documented disease

  * No tumor marker elevation as sole evidence of disease
* No necrotic/hemorrhagic metastases or tumor
* No untreated brain or meningeal metastases

  * Previously treated, radiologic or clinical evidence of stable brain metastases allowed provided disease is asymptomatic and corticosteroids are not required

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Hemoglobin normal
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN) OR creatinine clearance ≥ 50 mL/min
* Bilirubin ≤ 1.5 times ULN
* AST or ALT ≤ 2 times ULN (5 times ULN if liver involvement)
* Proteinuria ≤ grade 1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of other malignancies except adequately treated nonmelanoma skin cancer or other solid tumors curatively treated with no evidence of disease for ≥ 5 years
* No untreated and/or uncontrolled cardiovascular conditions or symptomatic cardiac dysfunction
* No resting blood pressure (BP) consistently higher than systolic BP > 150 mm Hg and diastolic BP > 100 mm Hg (in the presence or absence of a stable dose of antihypertensive medication)
* No poorly controlled hypertension, history of labile hypertension, or poor compliance with antihypertensive medication
* No overt bleeding (≥ 30 mL bleeding/episode) within the past 3 months
* No clinically relevant hemoptysis (≥ 5 mL fresh blood) within the past 4 weeks

  * Flecks of blood in sputum allowed
* No active or uncontrolled infections
* No serious illnesses or medical conditions that would preclude compliance with study requirements
* No mean QTc with Bazett's correction > 470 msec
* No history of familial long QT syndrome
* No peripheral neuropathy > grade 1
* No dihydropyrimidine dehydrogenase deficiency or history of severe hand-foot syndrome after fluoropyrimidines (for patients with CRC)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* At least 6 months since prior adjuvant or neoadjuvant therapy
* At least 6 months since prior adjuvant radiotherapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin C) (for patients with NSCLC)
* At least 4 weeks since prior and no concurrent corticosteroids
* At least 3 weeks since prior palliative radiotherapy and recovered

  * Concurrent palliative radiotherapy allowed
* At least 2 weeks since prior epidermal growth factor receptor inhibitor therapy
* At least 2 weeks since prior major surgery
* No more than 1 prior single-agent, nonplatinum-containing chemotherapy regimen for metastatic disease (for patients with NSCLC)
* No prior gemcitabine hydrochloride (for patients with NSCLC)
* No prior oxaliplatin (for patients with CRC)
* No prior angiogenesis inhibitor
* No prior chemotherapy for advanced/metastatic disease (for patients with CRC)
* No other concurrent experimental drugs or anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-11-29 (Actual); Primary Completion 2007-09-18 (Actual); Study Completion 2008-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Batist, MD, Study Chair — Jewish General Hospital; Eric X. Chen, MD, PhD, Study Chair — Princess Margaret Hospital, Canada; Glenwood D. Goss, MD, BCh, FCP, FRCPC, Study Chair — Ottawa Regional Cancer Centre
Locations (3):
- Canada (3):
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital - Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen E, Jonker D, Gauthier I, MacLean M, Wells J, Powers J, Seymour L. Phase I study of cediranib in combination with oxaliplatin and infusional 5-Fluorouracil in patients with advanced colorectal cancer. Clin Cancer Res. 2009 Feb 15;15(4):1481-6. doi: 10.1158/1078-0432.CCR-08-0761. PMID 19228749